CLINICAL TRIAL: NCT00672802
Title: A Phase II Safety Study of TAK-375 in Subjects With Mild to Moderate Chronic Obstructive Pulmonary Disease
Brief Title: Safety of Ramelteon in Subjects With Mild to Moderate Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-03-TL-375-038; U1111-1115-1343 (Registry Identifier: WHO)
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Insomnia; Drug Therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Initiation and Maintenance Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ramelteon 16 mg QD and Placebo QD (Experimental)
  Interventions: Drug: Ramelteon and Placebo

INTERVENTIONS:
Drug: Ramelteon and Placebo — Ramelteon 16 mg, tablet, orally, once daily for Periods 1 or 2 and ramelteon placebo-matching tablets, orally, once daily for Periods 1 or 2.
  Other Names: Rozerem™; ramelteon; TAK-375

SUMMARY:
This purpose of this study is to assess the safety of ramelteon, once daily (QD), in subjects with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Insomnia is characterized by difficulties initiating and maintaining sleep, or complaints of non-restorative and non-refreshing sleep. Transient insomnia affects approximately one-third to one-half of the US population, based on the results of 2 surveys of representative samples of the adult US population conducted by the Gallup Organization in which respondents were asked if they had "ever had difficulty sleeping." Based on reports of "regular" or "frequent" sleep difficulty, results from the same studies suggest that approximately one-tenth of the US population experiences chronic insomnia. The ideal treatment for insomnia would reduce the latency to onset of sleep and increase total sleep time, without a negative impact on sleep architecture and without safety concerns or next-day effects.

Ramelteon is under global development by Takeda Chemical Industries, Ltd., for the treatment of transient and chronic insomnia and for the treatment of Circadian Rhythm Sleep Disorders.

This study is being conducted to assess the safety of ramelteon in subjects with chronic obstructive pulmonary disease. Participation in the study is anticipated to be about 1.5 months.

ELIGIBILITY:
Inclusion Criteria

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Clinical history of chronic obstructive pulmonary disease and a confirmatory diagnosis based on pulmonary function tests at screening.
* Moderate: forced expiratory volume in one second/ forced vital capacity less than 70% and forced expiratory volume 135-75% of predicted.
* Post-bronchodilator forced expiratory volume in one second change from baseline of less than 12%.
* Negative chest x-ray at screening, other than findings consistent with mild to moderate chronic obstructive pulmonary disease, within the last 6 months.
* Arterial oxygen saturation during sleep greater than 85% for at least 99% of the recording period, with no arterial oxygen saturation readings less than 80% as assessed by pulse oximetry at polysomnography screening.
* Arterial oxygen saturation during wakefulness greater than 91% (both supine and sitting) as assessed by pulse oximetry at screening.
* Habitual bedtime is between 8:30 p.m. and 12:00 a.m.
* Body mass index between 18 and 34, inclusive.
* Agrees to remain in the study center for three overnight stays.

Exclusion Criteria:

* Known hypersensitivity to ramelteon or related compounds, including melatonin.
* Known hypersensitivity to Ventolin® or related compounds.
* Previously participated in a study involving ramelteon.
* Participated in any other investigational study and/or taken any investigational drug within 30 days or five half-lives prior to Day 1 of study medication, whichever is longer.
* Clinical history of acute or chronic respiratory failure, severe chronic obstructive pulmonary disease, or hypercapnia (Partial Pressure of Oxygen in Arterial Blood greater than or equal to45 mmHg).
* History of or currently has right ventricular hypertrophy on electrocardiogram or right heart failure.
* Periodic leg movement with arousal index (per hour of sleep) greater than 20 as seen at polysomnography screening.
* Apnea hypopnea index greater than 15 as seen at polysomnography screening.
* Acute clinically significant illness within 2 weeks or has been hospitalized within 4 weeks of study participation.
* Sleep schedule changes required by employment within three months prior to Day 1 of study medication, or has flown across greater than three time zones within seven days prior to screening.
* Participated in a weight loss program or has substantially altered their exercise routine within 30 days prior to Day 1 of study medications.
* History of seizures, sleep apnea, restless leg syndrome, period limb movement disorder, other known sleep disorders, schizophrenia, bipolar disease, mental retardation, or cognitive disorder.
* History of psychiatric disorder within the past 12 months.
* History of drug addiction or drug abuse within the past 12 months.
* History of alcohol abuse within the past 12 months and/or regularly consumes 4 or more alcoholic drinks per day.
* Unable to discontinue the use of hypnotics for the duration of the study.
* Any clinically important abnormal finding, other than chronic obstructive pulmonary disease, as determined by medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator.
* Current significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematologic, or metabolic disease, unless currently controlled and stable with protocol-allowed medication 30 days prior to Day 1 of study medication.
* Hematocrit value greater than 55% at screening.
* Positive hepatitis panel.
* Any additional condition(s) that in the Investigator's opinion would:

  * affect sleep-wake function
  * prohibit the subject from completing the study
  * not be in the best interest of the subject
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication, including:

  * Anxiolytics
  * Hypnotics
  * Antidepressants
  * Anticonvulsants
  * Sedating H1 antihistamines
  * Systemic steroids
  * Decongestants
  * Over-the-counter and prescription stimulants
  * Over-the-counter and prescription diet aids
  * Central nervous system active drugs and narcotic analgesics
  * Lipophilic beta blockers
  * Melatonin
  * St. John's Wort
  * Kava-kava
  * Gingko biloba

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2003-08; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Mean Oxygen Saturation during sleep for the entire night. | Periods 1 and 2.

SECONDARY OUTCOMES:
Mean Oxygen Saturation for each hour of the night. | Periods 1 and 2.
Mean Oxygen Saturation for awake Time Sleep Stage. | Periods 1 and 2.
Mean Oxygen Saturation for Nonrapid Eye Movement Sleep Stage. | Periods 1 and 2.
Mean Oxygen Saturation for Rapid Eye Movement Sleep Stage. | Periods 1 and 2.
Percentage of night when arterial oxygen percent saturation was less than 85%. | Periods 1 and 2.
Percentage of night when arterial oxygen percent saturation was less than 90%. | Periods 1 and 2.
Apnea Hypopnea Index measured by respiratory inductance plethysmography (RIP). | Periods 1 and 2.
Latency to Persistent Sleep. | Periods 1 and 2.
Total Sleep Time. | Periods 1 and 2.
Sleep Efficiency. | Periods 1 and 2.
Wake Time after Persistent Sleep Onset. | Periods 1 and 2.
Number of Awakenings after Persistent Sleep Onset. | Periods 1 and 2.
Subjective Sleep Latency. | Periods 1 and 2.
Subjective Total Sleep Time. | Periods 1 and 2.
Subjective Sleep Quality. | Periods 1 and 2.
Subjective Awake Time. | Periods 1 and 2.
Subjective Number of Awakenings. | Periods 1 and 2.
Subjective Ease of Falling Back to Sleep. | Periods 1 and 2.
Subjective Level of Alertness. | Periods 1 and 2.
Subjective Ability to Concentrate. | Periods 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science, Study Director — Takeda
Locations (6):
- United States (6):
  - Birmingham, Alabama
  - Santa Monica, California
  - Miami Beach, Florida
  - Winter Park, Florida
  - Louisville, Kentucky
  - Cincinnati, Ohio

REFERENCES:
- [Background] Kryger M, Wang-Weigand S, Zhang J, Roth T. Effect of ramelteon, a selective MT(1)/MT (2)-receptor agonist, on respiration during sleep in mild to moderate COPD. Sleep Breath. 2008 Aug;12(3):243-50. doi: 10.1007/s11325-007-0156-4. PMID 18060441
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI